CLINICAL TRIAL: NCT01368770
Title: Stress-rest Single Photon-Emission Computed Tomography(SPECT)Compared to Coronary Computed Tomographic Angiography in the Initial Evaluation of Patients With Suspected Coronary Artery Disease-A Pilot Randomized Controlled Trial
Brief Title: Stress Testing Compared to Coronary Computed Tomographic Angiography in Patients With Suspected Coronary Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Centre Hospitalier Universitaire de Bab El Oued (Other); Hospital Italiano Garibaldi,Rosario ARGENTINA (Unknown); Pontificia Universidad Catolica de Chile (Other); Fu Wai Hospital, Beijing, China (Other); Instituto de Cardiologia,Bogota D.C. COLOMBIA (Unknown); Instituto de Cardiologia y Cirugia Cardiovascular,LA Habana CUBA (Unknown); University Hospital Ostrava (Other); Indian Institute of Public Health, India (Other); Università degli Studi di Brescia (Other); Universidad Nacional Autonoma de Mexico (Other); University Medical Centre Ljubljana (Other); Ankara University (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Dr Ganesan Karthikeyan, Additional Professor of Cardiology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Protocol version 1.1; CTRI/2010/091/001384 (Registry Identifier: Clinical Trial Registry of India)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronary CTA (Experimental): Coronary CTA using standard protocols
  Interventions: Other: Coronary CTA; Other: Stress MPI SPECT
- Stress MPI SPECT (Active Comparator): Stress-rest MPI SPECT using standard protocols
  Interventions: Other: Coronary CTA; Other: Stress MPI SPECT

INTERVENTIONS:
Other: Coronary CTA — Coronary CTA using standard protocols
Other: Stress MPI SPECT — Stress MPI using standard protocols

SUMMARY:
The use of coronary computed tomographic angiography(CTA)is rapidly increasing, but there is lack of data which supports their use in the initial evaluation of patients who are asymptomatic or mildly symptomatic. The hypothesis underlying this proposal is that the use of stress-rest myocardial perfusion imaging (MPI) as an initial test for the evaluation of asymptomatic or mildly symptomatic patients who are at intermediate risk of coronary events will result in less further non-invasive and invasive testing and result in reduced costs, without adversely affecting clinical outcomes in the short term.

DETAILED DESCRIPTION:
Recently coronary computed tomographic angiography (CTA) has become increasingly popular as a means of investigating asymptomatic or mildly symptomatic patients, instead of stress-rest myocardial perfusion imaging (MPI), despite the absence of long-term prognostic data. With its high negative predictive value, CTA has become useful for exclusion of CAD in patients with chest pain syndromes. However, the clinical management of a patient with an abnormal CTA is not well defined. Further, several caveats remain regarding the use of coronary CTA. Despite the anatomic data provided by CTA, it does not yield information regarding the functional consequences of the obstruction. Moreover, this technique may miss small vessel disease because of limited resolution and may not be useful in the presence of significant vessel calcium or coronary stents. Most importantly, there is no long-term data regarding the prognostic ability of coronary CTA in the initial evaluation of patients at intermediate risk of coronary events. An abnormal CTA result often leads to additional functional testing or invasive coronary angiography. The major drawback of performing two or more tests in tandem is that it greatly adds to cost that can be prohibitive in lower and middle income countries. Therefore, there is a need to determine if either stress MPI or CTA performed initially, results in meaningful differences in costs without adversely affecting clinical outcomes.

The primary objective of this pilot study is to compare the efficacy (in terms of reduced additional non-invasive or invasive testing) and costs of a strategy of initial stress-rest MPI, to a strategy of initial coronary CTA in the management of asymptomatic or mildly symptomatic patients who are at intermediate risk of coronary events (death or nonfatal MI) by the Framingham criteria.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients above 21 years who are mildly symptomatic (those in class II NYHA), who have an intermediate likelihood of CAD, or asymptomatic patients who are determined to be at intermediate or high risk of coronary events by the Framingham (ATP III) criteria

Exclusion Criteria:

* Patients with prior documented CAD (by angiography), MI, coronary stenting or bypass surgery
* Patients in class III or IV NYHA
* Patients with chronic renal impairment to the extent of precluding contrast injection
* Severe medical disease with limited expectancy of life
* Contra-indication or allergy to pharmacologic stress agents or contrast agents
* Patients with unstable cardiac rhythms (including persistent atrial fibrillation) which preclude good ECG gating
* Weight limitations due to scanner design
* Pregnant/ lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have additional non-invasive testing with another modality, or invasive coronary angiography within 6 months of the first test. | 6 months
  The primary objective is to compare the efficacy (in terms of reduced additional non-invasive or invasive testing) and costs (at 6 months) of a strategy of initial stress-rest MPI, to a strategy of initial coronary CTA in the management of asymptomatic patients at intermediate or high risk of coronary events by the Framingham criteria, or mildly symptomatic patients who are at intermediate likelihood of having CAD.
Costs of investigation and treatment in both groups | 6 months
  To compare costs between a strategy of initial stress-rest MPI with a strategy of initial coronary CTA in the management of asymptomatic patients at intermediate or high risk of coronary events by the Framingham criteria, or mildly symptomatic patients who are at intermediate likelihood of having CAD.

SECONDARY OUTCOMES:
Proportion of patients who have planned, elective invasive angiography, elective coronary revascularization, or MACE at 6 month and at 1-year follow up | 6 months and 1 year
  To compare these two strategies in terms of the incidence of planned coronary angiography, revascularization and adverse clinical outcomes at 1 year (death, nonfatal MI, recurrent ischemia or unplanned coronary revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesan Karthikeyan, MD,DM,MSc, Principal Investigator — All India Institute of Medical Sciences; Salah E Bouyoucef, Principal Investigator — Centre Hospitalier Universitaire de Bab El-Qued; Jorge Cachero, Principal Investigator — Hospital Italiano Garibaldi; Rodrigo J Fernández, Principal Investigator — Universidad Católica de Chile; Zuo X He, Principal Investigator — Fu Wai Hospital, Beijing, China; Claudia Teresa G Villamil, Principal Investigator — Instituto de Cardiologia; Amalia T Peix González, Principal Investigator — Instituto de Cardiologia y Cirugia Cardiovascular; Otakar Kraft, Principal Investigator — University Hospital; Niveditha Devasenapathy, Principal Investigator — Indian Institute of Public Health; Davide Farina, Principal Investigator — Universita di Brescia; Aloha Meave, Principal Investigator — Universidad Nacional Autonoma de Mexico; Barbara G Salobir, Principal Investigator — University Medical Centre; Borut Jug, Principal Investigator — University Medical Centre; Elgin Ozkan, Principal Investigator — Ankara University; Maurizio DONDI, Principal Investigator — International Atomic Energy Agency; Ravi KASHYAP, Principal Investigator — International Atomic Energy Agency; Diana PAEZ, Principal Investigator — International Atomic Energy Agency
Locations (1):
- Department of cardiology, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Karthikeyan G, Guzic Salobir B, Jug B, Devasenapathy N, Alexanderson E, Vitola J, Kraft O, Ozkan E, Sharma S, Purohit G, Dolenc Novak M, Meave A, Trevethan S, Cerci R, Zier S, Gotthardtova L, Jonszta T, Altin T, Soydal C, Patel C, Gulati G, Paez D, Dondi M, Kashyap R. Functional compared to anatomical imaging in the initial evaluation of patients with suspected coronary artery disease: An international, multi-center, randomized controlled trial (IAEA-SPECT/CTA study). J Nucl Cardiol. 2017 Apr;24(2):507-517. doi: 10.1007/s12350-016-0664-3. Epub 2016 Oct 28. PMID 27796852